CLINICAL TRIAL: NCT01944761
Title: The Neuro-protective Effects of Exercise in Children Treated With Cranial Radiation for Brain Tumors
Brief Title: The Neuro-protective Effects of Exercise in Children With Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Donald Mabbott, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000019124
Record Dates: First submitted 2013-08-15; First posted 2013-09-18 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor
Keywords: Pediatrics; Brain Tumor; Neuro-radiation; Exercise
MeSH Terms: conditions — Brain Neoplasms; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Training (Experimental): The 16 participants in this group will be quasi-randomized based on the order of recruitment to start the 12 week exercise intervention without delay (immediate condition).
  Interventions: Behavioral: Exercise Program
- Delayed Exercise Training (Experimental): The 16 participants in this group will be quasi-randomized based on the order of recruitment to start the 12 week exercise intervention after a 12 week no exercise training period (delayed condition).
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — Designed to improve cardio-respiratory fitness, the exercise program will be conducted for 12 weeks at a frequency of 3-4 sessions per week. Each exercise session will be conducted after school for a total duration of 90 minutes (group sessions) or 30 minutes (home-based sessions). Group session activities will include i) warm-up (i.e. walk/jog, games) [10 mins], ii) aerobic training/fitness games [30 mins], iii) organized sports [30 mins], iv) cool down (i.e. stretching, low intensity games) [10 mins] and v) snack and reward (15 mins).
  Participants in the Group setting had three 90-minute group sessions per week. Participants in the Combined setting had two 90-minute group sessions and two 30-minute individual home-based sessions per week.

SUMMARY:
The objectives of our proposed study are to (a) evaluate the feasibility of conducting a structured exercise program in children treated with cranial radiation for brain tumors, (b) test whether exercise results in improved thinking skills and emotional function, and (c) examine potential mechanisms of improved outcome, particularly recovery of white matter and grey matter.

DETAILED DESCRIPTION:
Brain tumors are the leading cause of death and disability from childhood disease in developed countries. With treatment advances over the last 25 years, survival rates have improved dramatically. However, survival is often achieved at considerable cost. Cranial radiation is frequently required for effective tumor control, and is associated with significant neuro-toxicity, including white matter damage and cognitive morbidity. In order to achieve the best possible outcome for survivors, and ultimately conquer the long-term consequences of this disease, new interventions must be developed to ameliorate the neuro-toxic effects experienced by children. radiation injury can now be used to guide the development of interventions designed to rescue neural tissue. Furthermore, various new agents and activities with potential to stimulate neuro-recovery are now available. The potential value of exercise for rescuing the brain from neuro-toxic effects, for instance, has recently been reported. Next, neuro-cognitive processes that are particularly sensitive to the effects of cranial radiation have been identified and can serve as behavioral assays to test the effectiveness of these new interventions. Finally, novel neuro-imaging tools are available to perform in vivo evaluations in order to delineate potential mechanisms of neuro-recovery. We intend to integrate these new research findings to develop and evaluate a physical exercise-based intervention targeted at rescuing brain tissue of children with brain tumors from the neuro-toxic impact of cranial radiation.

ELIGIBILITY:
Inclusion Criteria:

* Survivors will be included if they are between 7 and 17 years of age.
* Survivors will be included if they either declare English as their native language or have had at least two years of schooling in English at the time of their first assessment.
* Survivors must have been diagnosed with a hemispheric or posterior fossa tumor and been treated with cranial spinal radiation.
* Survivors no more than 10 years may have elapsed between diagnosis and time of study.
* Survivors with a shunt will be included in the study, but will need to be identified prior to study on-set to discuss any specific considerations for imaging and physical activity.

Exclusion Criteria:

* are younger than 7 years (the delivery of an intervention program to young children carries challenges that make it difficult to include in an initial feasibility grant) or older than 17 years
* require sedation for MRI imaging
* is claustrophobic
* have severe neurological/motor dysfunction that would preclude safe participation in an exercise program.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2011-02-03 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2015-03-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing an excercise intervention | At week 42-45
  We will look at several factors, including recruitment rate, exercise adherence rate, retention rate and participant/parent satisfaction to determine the feasability of this intervention

SECONDARY OUTCOMES:
Fitness | Baseline, once at week 26-29 and once at week 42-45
  Fitness will be measured using the volume of oxygen consumed while exercising at maximum capacity (VO2max) on a stationary bicycle.
Neuro-cognitive outcome | Baseline, once at week 26-29 and once at week 42-45
  Three neuro-cognitive processes important for cognitive development, and found to be sensitive to radiation injury, will be assessed. These measures of cognition include attention, information processing speed, and declarative memory.
Neural recovery (gliogenesis/neurogenesis) | Baseline, once at week 26-29 and once at week 42-45
  Changes in white matter integrity may occur as a result of gliogenesis and will be measured using Diffusion Tensor Imaging (DTI). Neurogenesis occurs primarily within the hippocampus, a structure important for learning a memory. Cerebral blood flow (CBF) has been demonstrated to be a potential surrogate imaging measure of neurogenesis. As such, we will use Arterial Spin Labeled (ASL) perfusion MRI to obtain estimates of CBF within the hippocampus.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mabbott, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szulc-Lerch KU, Timmons BW, Bouffet E, Laughlin S, de Medeiros CB, Skocic J, Lerch JP, Mabbott DJ. Repairing the brain with physical exercise: Cortical thickness and brain volume increases in long-term pediatric brain tumor survivors in response to a structured exercise intervention. Neuroimage Clin. 2018 Mar 5;18:972-985. doi: 10.1016/j.nicl.2018.02.021. eCollection 2018. PMID 29876282
- [Background] Piscione PJ, Bouffet E, Timmons B, Courneya KS, Tetzlaff D, Schneiderman JE, de Medeiros CB, Bartels U, Mabbott DJ. Exercise training improves physical function and fitness in long-term paediatric brain tumour survivors treated with cranial irradiation. Eur J Cancer. 2017 Jul;80:63-72. doi: 10.1016/j.ejca.2017.04.020. Epub 2017 May 25. PMID 28551430
- [Background] Riggs L, Piscione J, Laughlin S, Cunningham T, Timmons BW, Courneya KS, Bartels U, Skocic J, de Medeiros C, Liu F, Persadie N, Scheinemann K, Scantlebury N, Szulc KU, Bouffet E, Mabbott DJ. Exercise training for neural recovery in a restricted sample of pediatric brain tumor survivors: a controlled clinical trial with crossover of training versus no training. Neuro Oncol. 2017 Mar 1;19(3):440-450. doi: 10.1093/neuonc/now177. PMID 27555603
- [Background] Cox E, Bells S, Timmons BW, Laughlin S, Bouffet E, de Medeiros C, Beera K, Harasym D, Mabbott DJ. A controlled clinical crossover trial of exercise training to improve cognition and neural communication in pediatric brain tumor survivors. Clin Neurophysiol. 2020 Jul;131(7):1533-1547. doi: 10.1016/j.clinph.2020.03.027. Epub 2020 Apr 13. PMID 32403066
- [Derived] Baudou E, Ryan JL, Cox E, Nham L, Johnston K, Bouffet E, Bartels U, Timmons B, de Medeiros C, Mabbott DJ. Optimizing an exercise training program in pediatric brain tumour survivors: Does timing postradiotherapy matter? Neurooncol Pract. 2023 Sep 9;11(1):69-81. doi: 10.1093/nop/npad055. eCollection 2024 Feb. PMID 38222057